CLINICAL TRIAL: NCT06498752
Title: A Phase II Clinical Trial of Consolidation Therapy Guided by MRD Testing After Radical Radiotherapy for Esophageal Cancer
Brief Title: MRD-Guided Consolidation Therapy Following Definitive Radiotherapy in Esophageal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Hebei Medical University Fourth Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEIR 2
Record Dates: First submitted 2024-06-20; First posted 2024-07-12 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Esophageal Cancer
Keywords: Esophageal squamous cell carcinoma; Immune checkpoint inhibitor; immunotherapy; chemotherapy; radiotherapy; Minimal residual disease, MRD
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma; Neoplasm, Residual

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRD negative (No Intervention): Intervention name: regular review of MRD monitoring; Intervention description: thoracic and abdominal CT, Esophagography and MRD monitoring every 3 months for 2 years after completion of radiotherapy
- MRD positive (Experimental): Intervention name: PD-1 monoclonal antibody consolidation therapy;
  Interventions: Drug: PD-1 monoclonal antibody consolidation therapy

INTERVENTIONS:
Drug: PD-1 monoclonal antibody consolidation therapy — PD-1 monoclonal antibody-based consolidation therapy for 1 year after completion of radiotherapy (or combination chemotherapy up to 4 cycles if less than 4 cycles of chemotherapy). Specific dosing: PD-1 monoclonal antibody, 200mg every 3 weeks.
  Arms: MRD positive

SUMMARY:
To further validate the performance of the high-sensitivity MRD assay in patients with squamous esophageal cancer who have completed radical radiotherapy; to validate whether MRD-negative patients can maintain a good prognosis under regular follow-up; and to validate whether MRD-positive patients can improve their survival with consolidation therapy with PD-1 monotherapy.

DETAILED DESCRIPTION:
Esophageal cancer is one of the most common lethal tumours in the world and accounts for more than 50% of new cases in China. Definitive concurrent chemoradiotherapy is the standard treatment for unresectable locally advanced esophageal cancer, and the 5-year survival rate is only about 30%, but due to the lack of evidence, consolidation therapy has not been explicitly recommended in major guidelines.

In the CheckMate 577 study, patients who did not achieve pathological complete response (pCR) after surgery improved their survival through immunology consolidation therapy with PD-1 monotherapy, suggesting that patients who did not achieve clinical complete response (cCR) after radiotherapy may benefit from immunology consolidation therapy. This suggests that patients who do not have a clinical complete response (cCR) after radiotherapy are likely to benefit from immunology consolidation therapy. Patients with cCR after radiotherapy may achieve similar results to those achieved with radical surgery, and consolidation is probably not necessary.

However, existing clinical practice is unable to accurately determine the efficacy of radiotherapy in esophageal cancer, making risk-of-recurrence-guided stratified consolidation strategies difficult to achieve. Most of the ongoing radiotherapy-immunotherapy studies in esophageal cancer have been designed to treat all patients indiscriminately with immunology consolidation therapy, which may lead to over-treatment of cCR patients.

Therefore, there is an urgent need to find easily accessible and reliable biomarkers for the efficacy of radiotherapy in esophageal cancer, and to carry out prospective clinical studies as soon as possible, so as to optimize the strategy of consolidation therapy after radiotherapy in esophageal cancer. The high sensitivity of minimal residual disease (MRD) detection technology established by the researcher's team provides a prerequisite for this.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years, any gender
2. Histologically or cytologically confirmed squamous cell carcinoma of esophageal cancer. The initial clinical stage is I-VIa (2018 AJCC Cancer Staging Manual, 8th Edition) , primary unresectable oesophageal cancer
3. ECOG performance status <= 1.
4. No significant abnormality in laboratory routine indicators such as blood routine and liver and kidney function
5. Completed radical radiotherapy (dose 50-60Gy);
6. Received a systemic regimen of platinum in combination with paclitaxel or a 5-FU-based two-drug regimen with or without PD-1 monotherapy in accordance with the CSCO guidelines, and S-1 monotherapy in elderly patients;
7. Informed consent

Exclusion Criteria:

1. Patients with other cancer history except hypopharyngeal carcinoma in situ, non-malignant skin cancer and cervical carcinoma in situ.
2. Active infection currently exists, serious illness such as myocardial infarction in the 6 months prior to enrolment
3. History of autoimmune diseases
4. Participate in other clinical trials at present or within 4 weeks before enrollment;
5. Received systemic therapy (chemotherapy alone or chemotherapy combined with immunotherapy) for more than 4 cycles.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Median progression-free survival (PFS) | 36 month
  Median progression-free survival (PFS), was defined as the time from the end of radiotherapy to the first documented progressive disease (PD) per RECIST 1.1 as assessed by the investigator, or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
5-year overall survival | 60 month
  Overall survival was defined as the time from the end of radiotherapy to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. OS is reported for all participants of the Intent-To-Treat (ITT) population. The Kaplan-Meier method was used to calculated the 5-year survival probability.
Cancer specific survival | 60 month
  From the end of radiotherapy to death specifically attributed to esophageal cancer.
Incidence of radiotherapy and immunotherapy related toxicity | Through study completion, an average of 3 year
  Acute toxicity Rate, was defined as the frequency of toxicities related to the treatment, which arises during radiotherapy and within three month after the end of radiotherapy, according to National Cancer Institute Common Terminology Criteria for Adverse Event,Version 5.0 (CTC AE5.0). Late toxicity rate, was defined as the frequency of toxicities related to the treatment, which arises three month after the end of radiotherapy, according to National Cancer Institute Common Terminology Criteria for Adverse Event,Version 5.0 (CTC AE5.0).
Quality of life score(QOL) for swallowing function | 36 month
  Evluated by the score of the participants through The EORTC Quality of Life Questionnaire - Oesophageal Cancer Module (EORTC QLQ-OES18). The EORTC QLQ-OES18 is a disease-specific questionnaire developed and validated to address measurements specific to esophageal cancer and contains 18 items assessing symptoms of dysphagia, pain, reflux symptoms, eating restrictions, anxiety, dry mouth, taste, body image, and hair loss. All subscale items were scored using a four-point Likert scale with the following response choices: 1=not at all, 2=a little, 3=quite a bit, 4=very much. Raw scores for the subscales were standardized into a range of 0 to 100 by linear transformation, with higher symptom scores represent a higher ("worse") level of symptoms.
General Quality of life score(QOL) | 36 month
  Change From Baseline in the EORTC QLQ-C30 Subscale Scores in Participants. The score of the participants evaluated by The EORTC core quality of life questionnaire (QLQ-C30). The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the Global Health Status (GHS) question were scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores were standardized so that scores ranged from 0 to 100, with a higher score represents a higher response level. Thus a high score for a functional scale represents a high/healthy level of functioning.

OTHER OUTCOMES:
Circulating DNA as biomarkers for the predicting of efficacy | 36 months
  To explore the dynamic changes of circulating tumor DNA (the frequency of specific mutations by Next-generation sequencing Methodology) from baseline, before and after radiotherapy and their relationship with recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital, CAMS, Beijing, Beijing Municipality, China